CLINICAL TRIAL: NCT05620030
Title: Evaluation of the Standard Data Collected as Part of the Erlangen Protocol for the Treatment and Monitoring of Patients With Univentricular Heart Defects in Terms of the Fontan Procedure
Brief Title: Prospective Evaluation of Univentricular Hearts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 528_20 B
Record Dates: First submitted 2022-09-21; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-09

CONDITIONS: Univentricular Heart
MeSH Terms: conditions — Univentricular Heart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Univentricular Heart (Experimental): All patients with univentricular hearts
  Interventions: Other: Univentricular Heart

INTERVENTIONS:
Other: Univentricular Heart — Prevention of complications when discovered

SUMMARY:
Univentricular heart defects are among the most complex congenital malformations. The treatment of these patients usually includes 3 operations and accompanying diagnostics, some of which are invasive, within the first 3 to 4 years of life until the "fontan circulation" is established. Unfortunately, the group of patients with a univentricular cardiac malformation is also the group with the highest mortality rate until the Fontan circulation is established. The expected mortality varies depending on the complexity of the underlying intracardiac and extracardiac malformations and possible concomitant morbidity; According to data from the National Quality Assurance in Germany, it is currently up to 30% in patients with hypoplastic left heart syndrome. However, the treatment methods are well standardized and there has been a clinical protocol in Erlangen since 2008 that includes diagnostic examinations using cardiac catheterization (HKU) and magnetic resonance imaging (MRT), as well as non-invasive, instrument-based diagnostics and targeted blood tests in a consistent sequence before and after the operations regulates. The Erlangen protocol ends with the cardiac MRT six months after the Fontan operation (syn: total cavopulmonary connection [TCPC]). If MRT imaging is not possible (e.g. if a cardiac pacemaker is present) or if there is a clinical indication (e.g. an obstruction noticeable on MRT or the presence of an "overflow with right-left shunt"), HKU is performed in the first year after TCPC. These examinations are used to depict hemodynamics, cardiac function, vascular development, and lymphatic drainage disorders in order to evaluate the preoperative risk, adapt treatment strategies to the individual, and identify complications at an early stage. This concept is based on clinical experience and current scientific findings and has proven itself in everyday clinical practice since its introduction for Erlangen-Fontan patients and has proven to be very helpful for individualized treatment. After a successful Fontan operation, the mortality risk in childhood is only low. In the long term, however, some of the patients unfortunately suffer from Fontan-typical long-term complications with protein-loss enteropathy having to be mentioned in particular, which is described in the literature with an incidence of 3-14% and today still a 5-year incidence-has a mortality risk of 6-12%.

DETAILED DESCRIPTION:
Univentricular heart defects are among the most complex congenital malformations. The treatment of these patients usually includes 3 operations and accompanying diagnostics, some of which are invasive, within the first 3 to 4 years of life until the "fontan circulation" is established. Unfortunately, the group of patients with a univentricular cardiac malformation is also the group with the highest mortality rate until the Fontan circulation is established. The expected mortality varies depending on the complexity of the underlying intracardiac and extracardiac malformations and possible concomitant morbidity; According to data from the National Quality Assurance in Germany, it is currently up to 30% in patients with hypoplastic left heart syndrome. However, the treatment methods are well standardized and there has been a clinical protocol in Erlangen since 2008 that includes diagnostic examinations using cardiac catheterization (HKU) and magnetic resonance imaging (MRT), as well as non-invasive, instrument-based diagnostics and targeted blood tests in a consistent sequence before and after the operations regulates. The Erlangen protocol ends with the cardiac MRT six months after the Fontan operation (syn: total cavopulmonary connection [TCPC]). If MRT imaging is not possible (e.g. if a cardiac pacemaker is present) or if there is a clinical indication (e.g. an obstruction noticeable on MRT or the presence of an "overflow with right-left shunt"), HKU is performed in the first year after TCPC. These examinations are used to depict hemodynamics, cardiac function, vascular development, and lymphatic drainage disorders in order to evaluate the preoperative risk, adapt treatment strategies to the individual, and identify complications at an early stage. This concept is based on clinical experience and current scientific findings and has proven itself in everyday clinical practice since its introduction for Erlangen-Fontan patients and has proven to be very helpful for individualized treatment.

ELIGIBILITY:
Inclusion Criteria:

* congenital heart defect of the univentricular type and the clinical necessity of a multi-stage treatment in terms of the Fontan procedure.

Exclusion Criteria:

* no exclusion criteria

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2031-05-20 (Estimated); Study Completion 2041-05-20 (Estimated)

PRIMARY OUTCOMES:
Number of correct findings in patients after Fontan palliation to assess the outcome after TCPC | 50 years
  correct perioperative course after TCPC, correct anatomy after surgery without vascular or anastomotic obstructions, correct cardiovascular function, correct lymphatic vessel presentation, correct liver sonography, blood protein values in the normal range, absence of clinical symptoms
Heart or valvular insufficiency assessed by echocardiography and MRI | 50 years
  Measured through ejaction fraction (EF; [EF]=%) and through visual assessment of the valves with e.g. doppler echocardiography.
  Additionally, measurement of the same values is performed through MRI
Pathologic presentation of lymph vessels assessed by MRI | 50 years
  Described through various scores (Biko et al., Schröder et al.)
Hypoalbuminemia, hypoproteinemia | 50 years
  measured through blood analysis (in g/L)
Number of patients with Protein-losing enteropathy (PLE) or plastic bronchitis | 50 years
  Assessed by clinical diagnosis
Number of patients with "Failing Fontan" | 50 years
  Examples would be Fontan take-down, heart transplant or passing away
Prevalence and cause of early post-Fontan morbidity | 50 years
  assessed by clinical diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Sven Dittrich, Prof., Study Chair — Universitätsklinikum Erlangen
Locations (1):
- Universitätsklinikum, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No